CLINICAL TRIAL: NCT04239547
Title: Effects of Recruitment Maneuver on Perioperative Pulmonary Complications in Hysterectomies
Brief Title: Effects of Recruitment Maneuver During Intraoperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Ozlem Sagir, MD, Associated professor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: osagir-4
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Laparoscopic Hysterectomy
Keywords: recruitment; pulmonary complication; oxygenisation
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Intervention Model Description: Group 1, Alveolar Recruitment Maneuver+positive end expiratory pressure (PEEP) Group 2, PEEP
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator, the participant and outcomes assessor will be masked to the intervention. Only the caregiver will be aware of the group and intervention received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recruitment (Experimental): Patients classified to receive recruitment maneuver + 5 mmHg positive end-expiratory pressure after anesthesia induction and intubation.
  Interventions: Procedure: Alveolar Recruitment maneuver (ARM) +PEEP
- Non-recruitment (Experimental): Patients classified to receive only 5 mmHg positive end-expiratory pressure after anesthesia induction and intubation.
  Interventions: Procedure: PEEP

INTERVENTIONS:
Procedure: Alveolar Recruitment maneuver (ARM) +PEEP — Following anesthesia induction and intubation, alveolar recruitment maneuver followed by 5 mmHg PEEP
  Arms: Recruitment
Procedure: PEEP — Following anesthesia induction and intubation, only 5 mmHg PEEP
  Arms: Non-recruitment

SUMMARY:
The aim of this study is to observe the effect of respiratory recruitment maneuver on intraoperative ventilatory parameters and postoperative pulmonary complications in patients over 18 years scheduled for laparoscopic hysterectomy.

DETAILED DESCRIPTION:
In patients over 18 years who are scheduled for laparoscopic hysterectomy volunteering to participate in our study will receive anesthesia induction with one of our standard general anesthesia protocols. After intubation recruitment maneuver will be applied to the study group. General anesthesia and mechanical ventilation will be continued and completed according to our standard practice without any further intervention. Throughout the intraoperative period respiratory and haemodynamic parameters including compliance, airway resistance, mean arterial pressure, heart rate, pulse oxymetry, blood gas analysis, the applied inhalational anesthetic agent, minimum alveolar concentration, expiratory agent concentration and total agent consumption will be recorded. At the end of the operation anesthesia will be terminated and patients will be transferred to postanesthesia care unit (recovery unit after recovery and further discharged from to the ward when their Aldrete score is >8. The patients will be examined for respiratory complications on postoperative day 1, and will be followed up by telephone on day 5.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I-II
* > 18 y
* laparoscopic hysterectomy patients

Exclusion Criteria:

* Patient refusal to participate in the study
* <18 y, BMI> 40
* Patients receiving invasive MV support in the last 1 month
* Patients who received chemotherapy or radiotherapy in the last 2 months
* Patients with severe pulmonary disease (COPD, asthma, pulm infection, bronchiectasis) (those who have previously received Non-Invasive MV, oxygen therapy or steroid therapy for an acute attack)
* Those with known severe pulmonary Hypertension
* Intracranial tm
* Hemodynamic instability
* Shock.
* Neuromuscular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
measurement of change in airway compliance | T1:1minute(min)after intubationT2:5 min after Mechanical Ventilation(MV),T3:5 min after pneumoperitoneum,T4:3 min after Trendelenburg position(TP),T5:10 min after TP T6:20 min after TP T7:10 min after pneumoperitoneum deflation T8:1 min before extubation
  the patients airway compliance will be monitorised as milliliter / centimeter of water (mL/cmH2O) continuously by the anesthesia machine and will be recorded intermittently.
measurement of change in Airway resistance | T1:1 minute after intubationT2:5 min after MV T3:5 minute after pneumoperitoneum T4:3 minute after Trendelenburg position (TP) T5:10 minutes after TP T6:20 minutes after TP T7:10 minutes after pneumoperitoneum deflation T8:1 minute before extubation
  the patients airway compliance will be monitorised as centimeter of water/ liter/ minute (cmH2O/L/min) continuously by the anesthesia machine and will be recorded intermittently.
measurement of change in partial oxygen pressure (PaO2) | T1:1 minute after intubation T7: 10 minute after pneumoperitoneum deflation
  Arterial blood samples will be obtained and analysed. PaO2 will be recorded from these samples.

SECONDARY OUTCOMES:
Evaluation of Postoperative respiratory distress, cough, phlegm | T9: 24 hours after surgery . T10: on postoperative day 5
  Pulmonary complications including respiratory distress, cough, phlegm will be evaluated by questionnaire and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University, Balıkesir, Turkey (Türkiye)